CLINICAL TRIAL: NCT05230602
Title: Can a Daily Consuming of Opuntia (Tzabar Fruit) Reduce Symptoms of Fatigue, Pain and Depression Among Women With Fibromyalgia
Brief Title: Consuming of Opuntia Among Women With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Orli Grinstein-Cohen PhD, Head of the Nursing Department Ben Gurion University, Soroka University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0207-21-SOR
Record Dates: First submitted 2021-12-14; First posted 2022-02-09 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Fibromyalgia (FM)
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: At the start of the study (T1), the participants will fill the above scales. The participants will then be divided randomly into two equal groups. Group A will be instructed to eat the tzabar fruit twice a day for two weeks, while Group B, the control group, will be instructed not to change their diet. At the end of 14 days (T2) all participants will be re-assessed again. Then Group B will be instructed to eat the tzabar fruit twice a day for 14 days, while Group A, will be instructed to eat their regular diet. During the research period, the participants will be instructed to continue their regular treatment routine, whether this includes taking medication, performing sporting activity, and so on in order to avoid undesirable influences that could bias the research results. The tzabar fruits will be supplied by the research team, in a neutral location. After a month all participants will fill the above scales.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The participants will fill the study scales and will be instructed to eat the tzabar fruit twice a day for two weeks
  Interventions: Dietary Supplement: opuntia (tzabar fruit)
- Control Group (No Intervention): The participants will fill the study scales and will be instructed not to change their diet for two weeks

INTERVENTIONS:
Dietary Supplement: opuntia (tzabar fruit) — consuming of the tzabar fruit twice a day
  Arms: Study Group

SUMMARY:
To examine whether the addition of tzabar fruit twice a day to a routine daily nutrition regime will:

A- Reduce symptoms of fatigue, pain and depression in FM patients

B. Have positive influence on quality of life

DETAILED DESCRIPTION:
Project description Fibromyalgia (FM) is a chronic and idiopathic syndrome, characterized by a general distributed pain, more prevalent in women. Alongside with musculoskeletal pain, symptoms of fatigue, depression, anxiety and cognitive dysfunction are reported by the patients .The underlying pathophysiology of FM is still poorly understood, and treatment is often unsatisfactory. Current research provides evidence for altered pain processing in chronic pain patients, and specifically in FM patients.

Treatment for this syndrome is challenging and focuses on alleviation of symptoms. Patients use prescribed medication together with different complementary and alternative medicine treatments. Yet, the lack of adherence to the established treatment is quite common. Some patients do not conform to prescribed medication and reduce the recommended dose or interrupt the treatment whereas others use overdoses and self-medication. It is important to note that the patient's quality of life was higher in patients with higher adherence to treatment and persistence. Due to the lack of specific and standardized treatments for the management of FM, available evidence suggests a multidisciplinary approach, and nutrition represents an important therapeutic strategy.

The rationale for the current study is based on the platform of other chronic disease and the beneficial effect of consuming opuntia fruits (tzabar). The investigators propose a change in diet to reduce fatigue and chronic pain.

The mechanism explaining the benefits of opuntia fruit-tzabar, are not fully clear. Yet, several proposed pathways are suggested in the literature. The effect of tzabar was studied in in vitro model by Nunes et al. (2011) using intestinal cells taken from patients with Crohn and Colitis. Nunes et al. (2011) found that tzabar extract reduced pro-inflammatory mediators' secretion of IL-8. The reduction of IL-8 was explained via the reduction of NFkB pathway activation. This pathway inhibits the nuclear translocation of the redox sensitive transcription factor NFkB. Another possible mechanism for alleviation of pain symptoms is the high percentages of polysaccharides that tzabar fruits contain. High levels of polysaccharides were related to inhibition of alpha glucosidase inhibitor through a barrier function. Furthermore, tzabar has high level of fibers such as pectin which are beneficial to a healthy diet regime.

The investigators will examine whether an addition of tzabar twice a day to a daily nutrition regime will reduce the symptoms of fatigue and pain among patients with FM.

Aims

1. To examine whether the consumption of tzabar fruit has a positive influence on the reduction of fatigue, pain and depressive symptoms among patients with FM.
2. To examine whether the consumption of tzabar fruit has a positive influence on quality of life of patients with FM.

Hypotheses

1. The consumption of tzabar fruit twice a day for one month will reduce symptoms of a) fatigue, b) pain and c) depression among patients with FM.
2. The consumption tzabar fruit twice a day for one month will have a beneficial influence on the quality of life of FM patients.

Method Longitudinal study design. Inclusion criteria are women diagnosed with FM, age over 18, fluent in Hebrew. Non-inclusion criteria are FM patients with known sensitivity to tzabar/exotic fruits, FM patients known to suffer from digestive issues, such as irritable bowel syndrome, FM patients participating in another interventional study. Removal criteria are participants who do not complete the study follow-up period. The patients will be recruited from the rheumatological clinic at the Soroka Medical Center. Each patient arriving at the clinic and answering the inclusion criteria will be invited to participate and will sign an informed consent. The clinic operated once a week. Patients arriving on even dates during the first month of the study will be entered to the study group whereas patients on odd dates will comprise the control group.

The investigators performed calculations to estimate sample size. The investigators expected a modest (2.9 points on a 10-point scale) reduction in pain, relative to control. Given previously reported SDs of 3.5 on this scale in fibromyalgia, following Rasmussen et al. (2012) the sample size needed to detect an effect of this size, with a two-tailed alpha of 0.05 and power of 0.80, was 15 per group.

Measurement Dependent variables (quality of life, anxiety, pain, fatigue, depression) will be measured using the Widespread Pain Index (WPI), and the Symptom Severity Scale (SSS), along with Hebrew version of the quality-of-life questionnaire SF-36. Depression will be assessed by Beck Depression Inventory. Those that will be detected with depression will be refer back to Dr. Zeler for advice and treatment. If needed the psychiatric ward will be informed to build treatment program.

Process At the start of the study (T1), the participants will fill the above scales. The participants will then be divided randomly into two equal groups. Group A will be instructed to eat the tzabar fruit twice a day for two weeks, while Group B, the control group, will be instructed not to change their diet. At the end of 14 days (T2) all participants will be re-assessed again. Then Group B will be instructed to eat the tzabar fruit twice a day for 14 days, while Group A, will be instructed to eat their regular diet. During the research period, the participants will be instructed to continue their regular treatment routine, whether this includes taking medication, performing sporting activity, and so on in order to avoid undesirable influences that could bias the research results. The tzabar fruits will be supplied by the research team, in a neutral location. After a month all participants will fill the above scales.

Statistical analysis of data The statistical analysis of the data will be conducted using SPSS software. Descriptive statistics will be employed to characterize the sample. The data will be presented as categorical, ordinal, or continuous variables. For categorical variables, the number of participants and the percentage in each category will be presented. Ordinal variables will be presented using the median and the frequent. Quantitative variables will be presented using the average and standard deviation values. The changes in QOL and fatigue measures in each study group during the follow-up period will be analyzed with two-way repeated measures ANOVA, and comparison between the group will be performed using MANOVA. Multivariate analysis will include General Linear Model (GLM) for each outcome. The independent variables will include the study group, study period, interaction variable (study group * period) and the baseline characteristics of the patients. The effect of mediation (SABRES - fatigue - QOL) will be analyzed with SOBEL test.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with FM
* Age over 18
* Fluent in Hebrew

Exclusion Criteria:

* sensitivity to tzabar/exotic fruits
* Suffer from digestive issues, such as irritable bowel syndrome
* Participating in another interventional study

Removal criteria

- Participants who do not complete the study follow-up period.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Fibromyalgia (FM) is a chronic and idiopathic syndrome, characterized by a general distributed pain, more prevalent in women
Enrollment: 19 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
consumption of tzabar fruit has a positive influence on the reduction of pain | Two weeks
  Pain will be measured using the Widespread Pain Index (WPI) higher scores indicate greater widespread pain
consumption of tzabar fruit has a positive influence on fatigue | Two weeks
  fatigue will be measured using the Symptom Severity Scale (SSS) (Wolfe et al.,2010). higher scores indicate severe Symptoms including fatigue
consumption of tzabar fruit has a positive influence on fatigue | Two weeks
  fatigue will be measured using the Hebrew version of the quality-of-life questionnaire SF-36 (Levin-Epstein et al., 1998) higher scores indicate beter QOL and less fatigue
consumption of tzabar fruit has a positive influence on depressive symptoms | Two weeks
  Depression will be assessed by Beck Depression Inventory (Beck, 1996). higher scores indicate severe depressive symptoms.Those that will be detected with depression will be refer back to the outpatient clinic for advice and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Orli Grinstein-Cohen, PhD, Principal Investigator — Ben-Gurion University of the Negev/Soroka Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Southern District, Israel

IPD SHARING:
Plan to Share IPD: No